CLINICAL TRIAL: NCT06710405
Title: The Effect of Intraoperative Intravenous Lidocaine Infusion on Postoperative Pain and Recovery in Children (< 7 Years Old) Undergoing Thoracoscopic Surgery:Prospective, Randomized Controlled Trial
Brief Title: The Effect of Intraoperative Intravenous Lidocaine Infusion on Postoperative Pain and Recovery in Children (< 7 Years Old) Undergoing Thoracoscopic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H2409-100-1573
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Pain Management After Surgery
Keywords: pediatric; thoracoscopic surgery; pain control; lidocaine
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine group (Experimental): Anesthesia induction is performed according to the standard protocol. Monitoring includes electrocardiography, pulse oximetry, arterial blood pressure, depth of anesthesia (Patient State Index, PSI), and pain score (Analgesia Nociception Index).
  In the lidocaine group, a single bolus dose of lidocaine 1.5 mg/kg is administered concurrently with the induction of anesthesia, followed by a continuous infusion of lidocaine at a rate of 1.5 mg/kg/hr.
  Interventions: Drug: Lidocaine (drug)
- Control group (Placebo Comparator): The control group receives a continuous infusion of normal saline in the same volume as that administered to the lidocaine group.
  Interventions: Drug: Saline infusion (placebo)

INTERVENTIONS:
Drug: Lidocaine (drug) — a single bolus dose of lidocaine 1.5 mg/kg is administered concurrently with the induction of anesthesia, followed by a continuous infusion of lidocaine at a rate of 1.5 mg/kg/hr.
  Arms: Lidocaine group
Drug: Saline infusion (placebo) — Continuous infusion of normal saline in the same volume as that administered to the lidocaine group.
  Arms: Control group

SUMMARY:
This study aims to investigate the efficacy of intraoperative intravenous lidocaine infusion on postoperative pain management and recovery in pediatric patients undergoing thoracoscopic pulmonary resection.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged under 7 years undergoing thoracoscopic pulmonary resection

Exclusion Criteria:

* cardiac dysfunction requiring vasopressors or inotropic agents
* atrioventricular block or bradycardia
* Liver or kidney dysfunction
* Hypersensitivity to local anesthetics

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FLACC (ace, Legs, Activity, Cry, Consolability scale) Score | up to 1 hour after surgery
  Highest FLACC Score recorded in the postanesthesia care unit (The scale is scored in a range of 0-10 with 0 representing no pain.)

SECONDARY OUTCOMES:
Remifentanil dose | throughout surgery (up to 3 hours)
  Total amount of remifentanil administered during surgery
ANI (Analgesia Nociception Index) | throughout surgery (up to 3 hours)
  ANI (Analgesia Nociception Index) values during surgery (scale ranging from 0 (indicating maximum pain) to 100 (indicating no pain))
FLACC scores | 6 hours, 12 hours, and 24 hours postoperatively
  FLACC scores at 6 hours, 12 hours, and 24 hours postoperatively
Total analgesic dosage administered postoperatively | up to 3 days after surgery
Postoperative complications | until discharge (up to 3-4 days after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided